CLINICAL TRIAL: NCT02993159
Title: Phase IIB Pre-Surgical Trial of Oral Tamoxifen Versus Transdermal 4-hydroxytamoxifen in Women With DCIS of the Breast
Brief Title: Testing an Active Form of Tamoxifen (4-hydroxytamoxifen) Delivered Through Breast Skin to Control Ductal Carcinoma in Situ (DCIS) of the Breast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); BHR Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCI 2015-06-04; P30CA060553 (NIH); NCI-2016-01911 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI 2015-06-04 (Other: Northwestern University); NWU2015-06-04 (Other: DCP); N01CN00035 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2016-12-15 (Estimated); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-09

CONDITIONS: Ductal Breast Carcinoma In Situ; Estrogen Receptor Positive
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — afimoxifene; 4,17 beta-dihydroxy-4-androstene-3-one; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (afimoxifene, placebo) (Experimental): Patients apply afimoxifene gel to both breasts and receive placebo PO daily for 4-10 weeks in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Afimoxifene; Other: Laboratory Biomarker Analysis; Other: Placebo
- Arm II (placebo, tamoxifen citrate) (Active Comparator): Patients apply placebo gel to both breasts and receive tamoxifen citrate orally PO daily for 4-10 weeks in the absence of disease progression or unexpected toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Drug: Tamoxifen Citrate

INTERVENTIONS:
Drug: Afimoxifene — Applied to the breast
  Other Names: 4-Hydroxy-Tamoxifen; 4-Hydroxytamoxifen; 4-OHT
  Arms: Arm I (afimoxifene, placebo)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm I (afimoxifene, placebo)
Other: Placebo — Applied to the breast
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo, tamoxifen citrate)
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI-46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide
  Arms: Arm II (placebo, tamoxifen citrate)

SUMMARY:
This randomized phase IIB trial studies how well tamoxifen or afimoxifene works in treating patients with estrogen receptor positive breast cancer. Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen citrate or afimoxifene may fight breast cancer by blocking the use of estrogen by the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that 2 mg once daily per breast of 4-hydroxytamoxifen (4-OHT) topical gel results in a reduction in the Ki-67 labeling index of ductal breast carcinoma in situ (DCIS) lesions that is not inferior to that seen with 20 mg daily oral tamoxifen citrate (TAM) for 4-10 weeks, when comparing the base-line diagnostic core biopsy to the therapeutic surgical excision sample.

SECONDARY OBJECTIVES:

I. To compare post-therapy changes in the oncotype DCIS-score between arms (this is a validated reverse transcriptase-polymerase chain reaction [RT-PCR] assay for Ki67, STK15, survivin, cyclin B1, MYBL2, PR, GSTM1).

II. To compare between-group post-therapy changes in immunohistochemistry (IHC) markers: CD-68 macrophage marker as a surrogate for response to therapy, p16 and COX-2.

III. To compare post-therapy changes in breast density, quantitative estimate, between arms.

IV. To compare post-therapy breast tissue and plasma levels of TAM and its metabolites (N-desmethyl tamoxifen [NDT], [E] and [Z] isomers of 4-hydroxytamoxifen [4-OHT], N-desmethyl-4-hydroxytamoxifen [endoxifen]).

V. To compare post-therapy breast tissue and plasma levels of estradiol and progesterone between arms (optional).

VI. To compare the post-therapy fraction of participants demonstrating "no residual DCIS".

VII. To compare post-therapy changes in plasma proteins involved in coagulation: factors VIII and IX, von Willebrand factor, total protein S between arms.

VIII. To compare post-therapy changes in plasma markers of systemic estrogenic effect (IGF-1, SHBG).

IX. To compare post-therapy changes in symptoms as captured in the breast cancer prevention trial (BCPT) Eight Symptom Scale (BESS) questionnaire and skin reactions to 4-OHT gel.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: Patients apply afimoxifene gel to both breasts and receive placebo orally (PO) daily for 4-10 weeks in the absence of disease progression or unexpected toxicity.

ARM II: Patients apply placebo gel to both breasts and receive tamoxifen citrate orally PO daily for 4-10 weeks in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up at 1-2 weeks and 1 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Screen-detected, estrogen receptor (ER) positive DCIS of the breast proven on core needle biopsy, defined as 10% positive cells; the presence of a focus suspicious for microinvasion will be allowed; the size of the DCIS in the core biopsy sample must total 5 mm (multiple cores can be summed) and must be estimated on the deepest step section (if step sections are taken)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Participants must have acceptable organ and marrow function as defined below:

Baseline lab parameters are not standard of care for initiation of tamoxifen therapy; a minimal panel will therefore be appropriate.

* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin within "≤1.5 x institutional upper limit of normal (ULN)institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal (ULN)
* Creatinine within "≤1.5 x institutional upper limit of normal (ULN) institutional limits
* Women of childbearing potential and their male partners must agree to use TWO effective forms of birth control (abstinence is not an allowed method) prior to study entry and for the duration of study participation, and for two months following the last dose of study medications; effective birth control methods are: copper IUD [intrauterine device], diaphragm/cervical cap/shield, spermicide, contraceptive sponge, condoms; women of childbearing potential must have a negative urine pregnancy test within seven days before starting study medications; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Willingness to avoid exposing breast skin to natural or artificial sunlight (i.e. tanning beds) for the duration of the study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* DCIS presentation as a palpable mass
* Exogenous sex steroid use within 4 weeks prior to core needle biopsy
* Prior ipsilateral breast cancer radiotherapy will be excluded; prior contralateral breast cancer therapy within 2 years will also be excluded
* Skin lesions on the breast that disrupt the stratum corneum (eg eczema, ulceration)
* History of endometrial neoplasia
* History of thromboembolic disease (history of varicose veins and superficial phlebitis is allowed)
* Current smokers
* Current users of potent inhibitors of tamoxifen metabolism must be able to discontinue their use and switch to an alternative medication for the duration of participation, under the advice of their physician; if the physician feels that an alternative medication is not appropriate for the subject and the current medication is medically necessary, the subject will not be eligible; the drugs are listed below; many of these are not in clinical use at the moment; bupropion, celecoxib, chlorpheniramine, chlorpromazine, cimetidine, citalopram, clemastine, clomipramine, clozapine, cocaine, delavirdine, desipramine, diphenhydramine, doxepin, duloxetine, escitalopram, fluoxetine, haloperidol, halofantrine, hydroxyzine, imipramine, isoniazid, ketoconazole, methadone, methimazole, mibefradil, miconazole, nicardipine, paroxetine, pergolide, perphenazine, pioglitazone, pyrimethamine, quinidine, quinine, ranitidine, ritonavir, ropinirole, sertraline, terbinafine, thioridazine, ticlopidine, tranylcypromine, trazodone, tripelennamine
* Prior use of SERMS or AIs including tamoxifen, raloxifene, anastrozole, letrozole, or exemestane for prevention or therapy within 5 years
* Participants may not be receiving any other investigational agents within 30 days of enrollment or during this study
* History of allergic reactions attributed to tamoxifen or compounds of similar chemical or biologic composition
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued by nursing mothers who agree to participate in the study
* Men are excluded from this study since DCIS of the breast is exceedingly rare in men, and there are no data regarding skin penetration of 4-OHT though male chest wall skin (which is thicker and hairier than female chest wall skin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, MD, Principal Investigator — Northwestern University
Locations (6):
- United States (6):
  - Northwestern University, Chicago, Illinois
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Khan SA, Mi X, Xu Y, Blanco LZ Jr, Akasha AM, Pilewskie M, Degnim AC, AlHilli Z, Amin AL, Hwang ES, Guenther JM, Kocherginsky M, Benante K, Zhang S, Helland T, Hustad SS, Gursel DB, Mellgren G, Dimond E, Perloff M, Heckman-Stoddard BM, Lee O. Presurgical Oral Tamoxifen vs Transdermal 4-Hydroxytamoxifen in Women With Ductal Carcinoma In Situ: A Randomized Clinical Trial. JAMA Surg. 2023 Dec 1;158(12):1265-1273. doi: 10.1001/jamasurg.2023.5113. PMID 37870954

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (4-OHT Topical Gel, Placebo): 2mg 4-hydroxytamoxifen (4-OHT) topical gel applied once daily per breast and placebo PO daily for 4-10 weeks
- Arm II (Placebo, Oral Tamoxifen): placebo gel applied once daily per breast and 20mg oral tamoxifen citrate PO daily for 4-10 weeks
Period: Overall Study
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Started | 47 | 53
Completed | 42 | 48
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Opted out of surgery | 2 | 0
Not completed — Surgery postponed due to COVID-19 and started AI | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Women with estrogen receptor positive DCIS
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen) | Total
Number analyzed (Participants) | 47 | 53 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 43 | 81
  >=65 years | 9 | 10 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 53 | 100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 42 | 45 | 87
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 7 | 19
  White | 31 | 34 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 47 | 53 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki-67 Labeling Index
Description: Change in the Ki-67 labelling index of DCIS lesions evaluated using immunohistochemistry
Time Frame: baseline to up to 10 weeks
Population: Participants with DCIS tissue samples at baseline and post-therapy
Measure: Mean (95% Confidence Interval); unit: percent positive cells
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 35 | 40
percent positive cells | -1.0 [-2.4 to 0.52] | -4.8 [-6.6 to -3.1]

2. Secondary Outcome: Change in Oncotype DCIS-Score
Description: Change in Exact Sciences Oncotype Diagnosis Breast Ductal Carcinoma in Situ Score (Oncotype DCIS-Score), a clinical validated clinically validated, commercially available genomic test for patients with DCIS. Oncotype DCIS-Score Range is 0-100. A negative change in scores indicates a lower risk of recurrence (better outcome).
Time Frame: baseline to up to 10 weeks
Population: Participants with Oncotype-DCIS score at baseline and post-therapy
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 32 | 28
score on a scale | -1.8 [-5.8 to 2.3] | -16 [-22 to -9.4]

3. Secondary Outcome: Post-therapy Breast Tissue Levels of Tamoxifen and Its Metabolites
Description: Post-therapy concentrations of 4-OHT and endoxifen in breast tissue samples
Time Frame: up to 10 weeks
Population: Participants with post-therapy tissue samples
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 40 | 47
ng/g
  4-OHT, Superficial tissue sample: number analyzed (Participants) | 36 | 43
  4-OHT, Superficial tissue sample | 4.2 [1.5 to 17.8] | 6.0 [3.9 to 8.5]
  4-OHT, Deep tissue sample: number analyzed (Participants) | 35 | 44
  4-OHT, Deep tissue sample | 3.8 [1.3 to 7.9] | 5.7 [4.0 to 7.9]
  Endoxifen, Superficial tissue sample: number analyzed (Participants) | 36 | 43
  Endoxifen, Superficial tissue sample | 0.2 [0.2 to 0.3] | 16 [9.5 to 20.7]
  4-OHT, Deep tissue sample: number analyzed (Participants) | 35 | 44
  4-OHT, Deep tissue sample | 0.3 [0.0 to 0.3] | 13 [8.9 to 20.6]

4. Secondary Outcome: Post-therapy Plasma Levels of Tamoxifen and Its Metabolites
Description: Post-therapy concentrations of 4-OHT and endoxifen in plasma samples
Time Frame: up to 10 weeks
Population: Participants with post-therapy plasma samples
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 39 | 47
ng/ml
  4-OHT, Plasma | 0.2 [0.1 to 0.4] | 2.0 [1.4 to 2.7]
  Endoxifen, Plasma | 0.0 [0.0 to 0.0] | 10.5 [6.4 to 13.8]

5. Secondary Outcome: Ki-67 Labelling Index in the Terminal Duct Lobular Units (TDLUs)
Description: Mean change in Ki-67 labelling index in the terminal duct lobular units (TDLUs)
Time Frame: baseline to up to 10 weeks
Population: Participants with terminal duct lobular units (TDLUs) at baseline and post-therapy
Measure: Mean (95% Confidence Interval); unit: percent positive
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 16 | 19
percent positive | -0.11 [-1.20 to 0.98] | 0.16 [-0.67 to 0.99]

6. Secondary Outcome: Change in Plasma Proteins Involved in Coagulation
Description: Mean change in percentage of plasma proteins involved in coagulation: Factor VIII, Factor IX, von Willebrand Factor, and total protein S
Time Frame: baseline to up to 10 weeks
Population: Participants with plasma samples at baseline and post-therapy
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 40 | 48
percent
  Factor VIII | -0.50 [-12 to 11] | -8.8 [-19 to 1.5]
  Factor IX | 0.07 [-7.4 to 7.6] | 2.2 [-2.0 to 6.4]
  vWF | 14 [-5.5 to 34] | 30 [16 to 44]
  Factor S | -2.9 [-7.7 to 1.9] | -11 [-17 to -4.9]

7. Secondary Outcome: Change in Plasma Markers of Systemic Estrogenic Effect (SHBG)
Description: Mean change in plasma markers of systemic estrogenic effect: SHBG.
Time Frame: baseline to up to 10 weeks
Population: Participants with plasma samples at baseline and post-therapy
Measure: Mean (95% Confidence Interval); unit: nmol/l
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 40 | 48
nmol/l | -0.24 [-10 to 9.9] | 15 [4.5 to 25]

8. Secondary Outcome: Change in Plasma Markers of Systemic Estrogenic Effect (IGF-1)
Description: Mean change in plasma markers of systemic estrogenic effect: IGF-1
Time Frame: baseline to up to 10 weeks
Population: Participants with plasma samples at baseline and post-therapy
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 40 | 48
ng/ml | -1.2 [-9.8 to 7.4] | -48 [-56 to -40]

9. Secondary Outcome: Change in Symptoms as Captured in the Breast Cancer Prevention Trial (BCPT) Eight Symptom Scale (BESS) Questionnaire and Skin Reactions to 4-OHT Gel.
Description: Mean change in symptoms as captured using the Breast Cancer Prevention Trial (BCPT) Eight Symptom Scale (BESS) questionnaire. A patient reported outcome, scores range from 0 (Not at All) to 4 (Extremely) when asked about experiencing symptoms. A positive change in scores indicates an increase in symptoms experienced and a negative change in scores indicates a decrease in symptoms experienced
Time Frame: baseline to up to 10 weeks
Population: Participants with BESS scores at baseline and post-therapy
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
Number analyzed (Participants) | 32 | 36
score on a scale
  Cognitive | 0.09 [-0.09 to .27] | -0.31 [-0.65 to 0.04]
  Body Pain | -0.10 [-0.33 to 0.12] | -0.15 [-0.37 to 0.08]
  Vasomotor | 0.15 [-0.08 to 0.37] | 0.53 [0.23 to 0.82]
  Gastrointestinal | -0.05 [-0.13 to 0.02] | -0.06 [-0.15 to 0.04]
  Sexual problems | 0.14 [-0.55 to 0.83] | -0.04 [-0.48 to 0.40]
  Bladder | -0.06 [-0.30 to 0.18] | -0.29 [-0.53 to -0.05]
  Body image | 0.04 [-0.03 to 0.11] | -0.04 [-0.12 to 0.04]
  Vaginal | -0.03 [-0.23 to 0.16] | -0.18 [-0.40 to 0.04]
  Problem | -0.01 [-0.06 to 0.04] | -0.04 [-0.11 to 0.04]

ADVERSE EVENTS:
Time Frame: up to 10 weeks
Arm/Group | Arm I (4-OHT Topical Gel, Placebo) | Arm II (Placebo, Oral Tamoxifen)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/53
Other Adverse Events (participants affected / at risk) | 27/47 | 33/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (4-OHT Topical Gel, Placebo) (N=47) | Arm II (Placebo, Oral Tamoxifen) (N=53)
Nausea (Gastrointestinal disorders) | 2 (47) | 6 (53)
Fatigue (General disorders) | 4 (4) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Breast Pain (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (9) | 8 (8)
Hot flashes (Vascular disorders) | 16 (18) | 21 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT02993159/Prot_SAP_ICF_000.pdf